CLINICAL TRIAL: NCT02732249
Title: A Randomized Clinical Trial of Clarithromycin/Bismuth Containing Quadruple Therapy for Helicobacter Pylori First-line Treatment
Brief Title: Clarithromycin Triple Therapy Plus Bismuth for Helicobacter Pylori First-line Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rjkls2016068
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Clarithromycin; Amoxicillin; Metronidazole; Eradication
MeSH Terms: interventions — Esomeprazole; Clarithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Triple regimen group (Active Comparator): Esomeprazole 20mg bid, clarithromycin 500mg bid and metronidazole 400mg qid for 14 days
  Interventions: Drug: Esomeprazole; Drug: Clarithromycin; Drug: Metronidazole
- Low metronidazole group (Experimental): Esomeprazole 20mg bid, bismuth potassium citrate 600mg bid, clarithromycin 500mg bid and metronidazole 400mg bid for 14 days
  Interventions: Drug: Esomeprazole; Drug: Bismuth Potassium Citrate; Drug: Clarithromycin; Drug: Metronidazole
- High metronidazole group (Experimental): Esomeprazole 20mg bid, bismuth potassium citrate 600mg bid, clarithromycin 500mg bid and metronidazole 400mg qid for 14 days
  Interventions: Drug: Esomeprazole; Drug: Bismuth Potassium Citrate; Drug: Clarithromycin; Drug: Metronidazole

INTERVENTIONS:
Drug: Esomeprazole — Given 30 min before morning and evening meals
Drug: Bismuth Potassium Citrate — Given 30 min before morning and evening meals
  Arms: High metronidazole group; Low metronidazole group
Drug: Clarithromycin — Given 30 min after morning and evening meals
Drug: Metronidazole — Given 30 min after meals or at bedtime

SUMMARY:
Standard triple therapy including a proton pump inhibitor (PPI) and clarithromycin with either amoxicillin or metronidazole are no longer recommended as empirical ﬁrst-line therapy to treat Helicobacter pylori infection because of high antibiotic resistance. It is unknown whether the addition of bismuth overcome antibiotic resistance. This study is designed to evaluate the efficacy and safety of the addition of bismuth to standard triple therapy for H. pylori first-line eradication.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-ulcer functional dyspepsia or scarred peptic ulcer disease
* Ability and willingness to participate in the study and to sign and give informed consent
* confirmed H. pylori infection

Exclusion Criteria:

* Previous H. pylori eradication therapy
* Less than 18 years old
* With history of H. pylori infection treatment
* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs
* Administration of antibiotics, bismuth, antisecretory drugs in 8 weeks prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy

SECONDARY OUTCOMES:
Rate of adverse effects | within 7 days after completion of therapy
Compliance rate | within 7 days after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hong lu, MD, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No